CLINICAL TRIAL: NCT03312621
Title: Implementing a Randomized Care Coordination Intervention for Minority Youth With Special Health Care Needs During Health Care Transition From Pediatric to Adult Health Care.
Brief Title: Improving Health Care Transition for Youth With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Tuchman (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Lisa Tuchman, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro2500; R40MC23627 (Other Grant/Funding Number: HRSA MCHB)
Record Dates: First submitted 2017-10-03; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Health Care Transition; Care Coordination
Keywords: Adolescent Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group received all aspects of enhanced usual care but was also assigned a healthcare transition nurse who coordinated the delivery of specific intervention services. These services included 1) a face-to-face systematic review of the readiness assessment with the participant/caregiver 2) a status assessment of ongoing healthcare transition planning and preparation; 3) monthly phone calls with the participant/caregiver to update and fill gaps in the healthcare transition action plan.
  Interventions: Behavioral: Health Care Transition Care Coordination
- Control (No Intervention): The control group received enhanced usual care which provides standardized healthcare transition-specific written information including a written transition policy, as well as insurance and guardianship information. Participants were also provided with a transition readiness assessment and entered into a healthcare transition registry to facilitate tracking and communication.

INTERVENTIONS:
Behavioral: Health Care Transition Care Coordination — These services included 1) a face-to-face systematic review of the readiness assessment with the participant/caregiver 2) a status assessment of ongoing healthcare transition planning and preparation; 3) monthly phone calls with the participant/caregiver to update and fill gaps in the healthcare transition action plan.
  Arms: Intervention

SUMMARY:
Special opportunities exist in vulnerable populations with chronic conditions to better understand what life course factors can facilitate attainment of optimal health and development. One such opportunity arises in the life of an adolescent or young adult when they transition their care from pediatric to adult health providers and systems, referred to as "health care transition". Experts generally agree that health care transition is often unsuccessful and associated with a variety of adverse outcomes. Adverse outcomes of unsuccessful health care transition include foregone or delayed medical care and having no identified adult medical home after leaving pediatrics. This foregone and delayed care can result in potentially preventable costly utilization of hospital emergency and inpatient services. Particularly concerning is increasing evidence that for some youth, transition from pediatric to adult medical care is a high-risk period for mortality. In addition to the adverse effects on individuals, unsuccessful health care transition also likely has economic consequences, particularly given that the majority of health care spending is already allotted to individuals with chronic conditions. These problems are even greater for low income and minority youth, with the District of Columbia having the highest level of unmet transition needs in the U.S.

DETAILED DESCRIPTION:
Special opportunities exist in vulnerable populations with chronic conditions to better understand what life course factors can facilitate attainment of optimal health and development. One such opportunity arises in the life of an adolescent or young adult when they transition their care from pediatric to adult health providers and systems, referred to as "health care transition". Experts generally agree that health care transition is often unsuccessful and associated with a variety of adverse outcomes. Adverse outcomes of unsuccessful health care transition include foregone or delayed medical care and having no identified adult medical home after leaving pediatrics. This foregone and delayed care can result in potentially preventable costly utilization of hospital emergency and inpatient services. Particularly concerning is increasing evidence that for some youth, transition from pediatric to adult medical care is a high-risk period for mortality. In addition to the adverse effects on individuals, unsuccessful health care transition also likely has economic consequences, particularly given that the majority of health care spending is already allotted to individuals with chronic conditions. These problems are even greater for low income and minority youth, with the District of Columbia having the highest level of unmet transition needs in the U.S.

In light of these facts, it becomes urgent to implement recommended standards for health care transition and evaluate their impact on transition outcomes. This research quantifies the impact of recommended health care transition practices using a randomized trial design and analysis following the intention-to-treat paradigm. The investigators do so by comparing aspects of 1) health care transition effectiveness (i.e., care coordination, timing, and services received); 2) experience of care (i.e., satisfaction and quality of chronic illness care); and 3) health care utilization in a population of 18-22 year-old African-American adolescents with special health care needs, receiving primary care in an urban academic adolescent medicine practice, using standardized outcome measures. Half of participants received usual care enhanced by written transition information, and half received a health care transition intervention modeled on the joint American Academy of Pediatrics, the American Academy of Family Physicians, and the American College of Physicians best practices report, released July 2011 that identified six recommended core components for transition programs. These include both practice based components (i.e. written transition policy, transitioning youth registry, and transfer of care) and patient level components (i.e. transition planning and completion). This report makes available an important standard for establishing transition practices but also demands careful evaluation.

ELIGIBILITY:
Inclusion Criteria:

* African-American, 16-22 years old at enrollment, receiving primary care at Adolescent Health Center, Recipient of Health Services for Children with Special Needs, Inc. insurance.

Exclusion Criteria:

* Exclusion criteria include individuals who have already been transferred from the adolescent health center to another practice and those with insufficient knowledge of English to participate in the telephone interviews.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 209 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Care Coordination | 2 years
  Mean score of Client Perceptions of Coordination Questionnaire (CPCQ)

SECONDARY OUTCOMES:
Patient-level experiences of care | 2 years
  Mean score of Patient Assessment of Chronic Illness Care Questionnaire (PACIC)
Healthcare utilization | 2 years
  Summary statistics of healthcare utilization
Healthcare cost | 2 years
  Summary statistics of healthcare cost

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K Tuchman, MD, MPH, Principal Investigator — Children's National Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lemke M, Kappel R, McCarter R, D'Angelo L, Tuchman LK. Perceptions of Health Care Transition Care Coordination in Patients With Chronic Illness. Pediatrics. 2018 May;141(5):e20173168. doi: 10.1542/peds.2017-3168. Epub 2018 Apr 12. PMID 29650807